CLINICAL TRIAL: NCT01130961
Title: Management of Advanced Non-Small Cell Lung Cancer and Clinical Outcomes in Patients Who Received Gefitinib (IRESSA) in Tertiary Care Setting in Thailand
Brief Title: Management of Advanced Non-Small Cell Lung Cancer (NSCLC) and Clinical Outcomes in Patients Who Received Gefitinib in Thailand
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-OTH-IRE-2009/1
Record Dates: First submitted 2010-04-29; First posted 2010-05-26 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Lung Cancer
Keywords: Advanced NSCLC; Gefitinib; Thai patient
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine progression-free survival of lung cancer patients who received gefitinib in clinical practice in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having lung cancer based on histological/cytological findings
* Admitted to the hospital between January 2004 and December 2008
* Treated with gefitinib for at least 3 months

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study
* Participation in another clinical study during the last 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lung cancer patients admitted in Chulalongkorn and Siriraj hospitals between January 2004 and December 2008 and treated with gefitinib for at least 3 months
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | median time from the first date of treatment until date of disease progression during Jan 2004- Dec 2008 or 5 years approx.

SECONDARY OUTCOMES:
Time to maximum response | Median time from the first date of treatment until the date that the disease can be maximum controlled during Jan 2004- Dec 2008 or 5 years approx.
Overall survival | time from the first date of treatment until date of patients dead during Jan 2004- Dec 2008 or 5 years approx.
Prevalence of EGFR & KRAS mutation from laboratory result | During Jan 2004- Dec 2008 or 5 years approx.

CONTACTS AND LOCATIONS:
Overall Officials: Virote Sriuranpong, MD., PhD., Principal Investigator — Chulalongkorn Hospital, Bangkok, Thailand; Vichien Srimuninnimit, MD., Principal Investigator — Siriraj Hospital, Bangkok, Thailand
Locations (1):
- Research Site, Bangkok, Thailand